CLINICAL TRIAL: NCT03991312
Title: A Two-Part, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Multiple Doses of Itraconazole and Rifampin on the Single-Dose Pharmacokinetics of Mitapivat Sulfate (AG-348) in Healthy Adult Subjects
Brief Title: Study to Evaluate the Effect of Multiple Doses of Itraconazole and Rifampin on the Single-Dose Pharmacokinetics of Mitapivat Sulfate (AG-348) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-012
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Itraconazole; Rifampin; mitapivat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Period 1: Day 1, participants will receive 20 milligrams (mg) of mitapivat sulfate.
  Period 2: Day 1 to Day 9, participants will receive 200 mg of itraconazole, once daily and 20 mg of mitapivat sulfate on Day 5.
  Interventions: Drug: itraconazole; Drug: mitapivat sulfate
- Part 2 (Experimental): Period 1: Day 1, participants will receive 50 milligrams (mg) of mitapivat sulfate.
  Period 2: Day 1 to Day 12, participants will receive 600 mg of rifampin, once daily and 50 mg of mitapivat sulfate on Day 8.
  Interventions: Drug: rifampin; Drug: mitapivat sulfate

INTERVENTIONS:
Drug: itraconazole — Participants will receive an oral solution as described in the arm description.
  Arms: Part 1
Drug: rifampin — Participants will receive oral capsule(s) as described in the arm description.
  Arms: Part 2
Drug: mitapivat sulfate — Participants will receive an oral tablet as described in the arm description.
  Other Names: AG348

SUMMARY:
Part 1 of this study will determine the effect of multiple-dose itraconazole, a strong cytochrome P450 (CYP) 3A4 and P-glycoprotein (P-gp) inhibitor, on the single-dose pharmacokinetic(s) (PK) of mitapivat sulfate in healthy adult participants. Part 2 of this study will determine the effect of multiple-dose rifampin, a strong CYP3A4 and P-gp inducer, on the single-dose pharmacokinetic(s) (PK) of mitapivat sulfate in healthy adult participants.

DETAILED DESCRIPTION:
This study consists of 2 periods and 2 parts. Participants will be placed in Part 1 or Part 2, and cannot participate in both:

Part 1, Period 1 includes a screening period up to 28 days prior to dosing and treatment on Day 1.

Part 1, Period 2 includes a treatment period from Day 1 to Day 9 and a possible follow-up, up to 28 days after the last dose of study drug.

Part 2, Period 1 includes a screening period up to 28 days prior to dosing and treatment on Day 1.

Part 2, Period 2 includes a treatment period from Day 1 to Day 12 and a possible follow-up, up to 28 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (non-childbearing potential), 18-55 years of age, inclusive, at the time of providing written informed consent;
* Continuous non-smoker who has not used nicotine-containing products for at least 12 months prior to screening, based on participant self-reporting, and agrees to abstain from use throughout the study;
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m2) at screening;
* Medically healthy, with no clinically significant conditions or abnormalities, as determined by the principal investigator (PI) or designee, through evaluation of medical history and screening vital signs, 12-lead electrocardiogram (ECG) results, physical examination findings, and clinical laboratory test results;
* A female participant must be of non-childbearing potential and must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

  * hysteroscopic sterilization;
  * bilateral tubal ligation or bilateral salpingectomy;
  * hysterectomy;
  * bilateral oophorectomy.
  * or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels at screening consistent with postmenopausal status;
* A male participant (with or without prior vasectomy) must agree to use a condom with spermicide or abstain from sexual intercourse from the time of providing written informed consent until 90 days after the last dose of study drug;
* If male, must agree not to donate sperm from the first dosing until 90 days after the last dose of study drug;
* Understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the study procedures and the protocol requirements, and has provided signed written informed consent prior to performing any study procedures, including screening procedures;

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study;
* History or presence of any clinically significant medical or psychiatric condition or disease or clinically significant laboratory abnormality that, in the opinion of the PI or designee, might confound the results of the study, compromise the ability of the participant to complete study procedures, and/or pose an additional risk to the participant by their participation in the study. This includes seizure disorders, transient ischemic attacks, or easy bruising;
* History or presence of a medical condition or surgical procedure that, in the opinion of the PI or designee, may potentially interfere with absorption, distribution, metabolism, or excretion of the study drugs;
* History or presence of alcohol or drug abuse within the past 2 years prior to screening;
* History or presence of hypersensitivity, idiosyncratic reaction, or serious adverse reaction to any of the study drugs or to their formulation excipients;
* Female participants of childbearing potential;
* Female participants with a positive serum pregnancy test at screening or check-in or who are breastfeeding;
* Positive urine drug or alcohol results at screening or check-in;
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody;
* Supine blood pressure is less than 90/40 milliliters of mercury (mmHg) or greater than 140/90 mmHg at screening. If the participant's systolic blood pressure reading exceeds 140 mmHg or the diastolic blood pressure reading exceeds 90 mmHg due to what may be, in the opinion of the PI or designee, an episode of transient anxiety, the reading may be repeated, and the resulting blood pressure measurement used to determine eligibility;
* Supine heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening. If the participant's heart rate exceeds 99 bpm due to what may be, in the opinion of the PI or designee, an episode of transient anxiety, the reading may be repeated, and the resulting heart rate measurement used to determine eligibility;
* QTcF interval is >450 milliseconds (msec) (males) or >470 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening;
* Estimated creatinine clearance < 90 mL/min at screening (Cockcroft-Gault formula);
* Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, proton pump inhibitors, H2-antagonists, herbal remedies, and vitamin supplements, beginning 28 days prior to the first dosing and throughout the study. Additionally, any drugs (with the exception of the study drugs) known to be clinically significant inhibitors or inducers of CYP3A, CYP2C9, CYP2C8, CYP2C19, and CYP1A2 enzymes and/or P-gp, including St. John's Wort, beginning 28 days prior to the first dosing and throughout the study. Appropriate sources (e.g., Flockhart TableTM) will be consulted to confirm lack of PK/PD interaction with study drugs. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee;
* Has consumed foods or beverages containing caffeine or xanthines 24 hours prior to the first dosing and is not willing to refrain from consumption of these foods or beverages throughout the study;
* Has consumed alcohol 48 hours prior to the first dosing and is not willing to refrain from consumption of alcohol throughout the study;
* Has consumed foods or beverages containing grapefruit or Seville oranges for 14 days prior to the first dosing and is not willing to refrain from consumption of these foods or beverages throughout the study;
* Has consumed fruit juices 72 hours prior to the first dosing and is not willing to refrain from consumption of these juices throughout the study
* Has consumed vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussel sprouts, and mustard), and charbroiled meats for 7 days prior to first dosing and is not willing to refrain from consumption of these foods throughout the study;
* Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing;
* Donation of blood or significant blood loss (≥500 mL) within 3 months prior to the first dosing and must be willing to refrain from voluntary blood donation for at least 30 days after the last dose of study drug;
* Plasma donation within 7 days prior to screening;
* Has liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin that are greater than the upper limit of normal at screening or check-in (confirmation of results may be done once);
* Has platelet, hemoglobin, and hematocrit that are below the lower limit of normal at screening or check-in (confirmation of results may be done once).
* History or presence of liver disease;
* Are currently enrolled in or have participated in another clinical study involving ongoing therapy with any investigational or marketed product or placebo within 3 months prior to the first dosing. The 3-month window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Treatment Period 1 of the current study;
* Has exposure to any investigational drug within 5 times the elimination half-life, if known (for marketed product) or within 3 months (if the elimination half-life is unknown) prior to first dosing;
* Has undergone any major surgical procedure within 3 months prior to Screening;
* History or presence of a primary malignancy, with the exception of a malignancy that has been curatively treated and for which the participant has displayed no evidence of disease within the 12 months prior to Screening;
* History or presence of a clinically significant allergy requiring medical treatment, as assessed by the PI or designee;
* Has glucose-6-phosphate dehydrogenase deficiency;
* Has veins that are unsuitable for multiple venipunctures/cannulation, as assessed by the PI or designee at screening;
* For Part 1 Only (Itraconazole):

  * History or presence of any of the following, deemed clinically significant by the PI or designee:

    * History or presence of ventricular dysfunction or risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, myocardial infarction, angina, unexplained syncope, personal or family history of Long QT Syndrome, Brugada syndrome, or sudden death).;
    * Uncorrected hypokalemia (potassium levels < 3.7) and/or hypomagnesemia (magnesium levels < 1.9).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve, from Time 0 to the Last Measurable Concentration (AUC0-t) of Mitapivat Sulfate with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Area Under the Concentration-Time Curve, from Time 0 to the Last Measurable Concentration (AUC0-t) of Mitapivat Sulfate with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of Mitapivat Sulfate with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of Mitapivat Sulfate with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Maximum Observed Plasma Concentration (Cmax) of Mitapivat Sulfate with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Maximum Observed Plasma Concentration (Cmax) of Mitapivat Sulfate with and without Rifampin | Predose and at various timepoints through 120 hours postdose

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve, from Time 0 to Hour 24 (AUC0-24) of Mitapivat Sulfate and AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Area Under the Concentration-Time Curve, from Time 0 to Hour 24 (AUC0-24) of Mitapivat Sulfate and AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Percent of AUC0-inf Extrapolated (AUC%extrap) of Mitapivat Sulfate and AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Percent of AUC0-inf Extrapolated (AUC%extrap) of Mitapivat Sulfate and AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Time of the Last Measurable Concentration (Tlast) of Mitapivat Sulfate and AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Time of the Last Measurable Concentration (Tlast) of Mitapivat Sulfate and AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Time to Reach Cmax (Tmax) of Mitapivat Sulfate and AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Time to Reach Cmax (Tmax) of Mitapivat Sulfate and AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Apparent First-Order Terminal Elimination Half-Life (t1/2) of Mitapivat Sulfate and AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Apparent First-Order Terminal Elimination Half-Life (t1/2) of Mitapivat Sulfate and AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Apparent Volume of Distribution During the Terminal Elimination Phase After Oral (Extravascular) Administration (Vz/F) of Mitapivat Sulfate with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Apparent Volume of Distribution During the Terminal Elimination Phase After Oral (Extravascular) Administration (Vz/F) of Mitapivat Sulfate with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Mitapivat Sulfate with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Mitapivat Sulfate with and without Rifampin | Predose and at various timepoints through 120 hours postdose
AUC0-t of AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
AUC0-t of AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
AUC0-inf of AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
AUC0-inf of AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Cmax of AGI-8702 with and without Itraconazole | Predose and at various timepoints through 120 hours postdose
Cmax of AGI-8702 with and without Rifampin | Predose and at various timepoints through 120 hours postdose
Percentage of Participants Experiencing an Adverse Event | Baseline up to a maximum of 38 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States